CLINICAL TRIAL: NCT03505021
Title: Effects of Oral Levosimendan (ODM-109) on Respiratory Function in Patients With ALS
Acronym: REFALS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Orion Corporation, Orion Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 3119002
Record Dates: First submitted 2018-04-16; First posted 2018-04-20 (Actual); Results first posted 2021-08-31 (Actual); Last update posted 2022-05-11 (Actual); Status verified 2022-04

CONDITIONS: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — Simendan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Levosimendan (Experimental): Levosimendan 1 mg capsules for oral administration, once to twice a day. The total duration of treatment 48 weeks
  Interventions: Drug: Levosimendan
- Placebo for levosimendan (Placebo Comparator): Placebo capsule for oral administration, once to twice a day. The total duration of treatment 48 weeks.
  Interventions: Drug: Placebo for levosimendan

INTERVENTIONS:
Drug: Levosimendan — Levosimendan 1 mg capsule for oral administration
  Other Names: ODM-109
  Arms: Levosimendan
Drug: Placebo for levosimendan — Placebo capsule for oral administration
  Other Names: Placebo for ODM-109
  Arms: Placebo for levosimendan

SUMMARY:
This study will evaluate whether prolonged oral levosimendan can preserve respiratory function more effectively than placebo, resulting in better patient functionality as measured by the ALSFRS-R scale. In this randomized, double-blind, placebo-controlled, parallel-group, multicenter study, subjects are allocated in a 2:1 ratio to receive either levosimendan (1 -2 mg daily) or placebo for 48 weeks. The primary endpoint is slow vital capacity (SVC) at 12 weeks, with the impact on patient function assessed through 48 weeks, adjusted for patient outcome, using ALSFRS-R (combined assessment of function and survival, CAFS). Other important efficacy measures include time to respiratory events, clinical global impression (CGI), assessment of dyspnea using the Borg scale and sleep scales (Pittsburgh sleep quality index and Epworth sleepiness scale). Patient safety is monitored using conventional methods including adverse events, safety laboratory tests, vital signs and 12-lead EKG. Following screening and baseline visits, patients attend the clinic at 2, 4, 8, 12, 24, 36 and 48 weeks, with telephone assessments conducted at weeks 18, 30 and 42. An end of study visit is performed 14-25 days after the last study treatment administration. The study will be monitored by an independent data and safety monitoring board. A long-term extension study will be available for patients completing the study.

ELIGIBILITY:
Inclusion Criteria:

* Written or verbal informed consent (IC) for participation in the study
* Male or female subjects with diagnosis of laboratory supported probable, probable or definite ALS according to El Escorial revised criteria. Full electromyogram (EMG) report available consistent with ALS (but not necessarily fulfilling the electrodiagnostic criteria for ALS) from an experienced neurophysiologist
* Able to swallow study treatment capsules, and in the opinion of the investigator, is expected to continue to do so during the study
* Sitting SVC between 60-90% of the predicted value for age, height and sex at screening visit
* Disease duration from symptom onset (defined by first muscle weakness or dysarthria) 12-48 months at the time of visit 1 (baseline)
* Able to perform supine SVC in an adequate and reliable way at screening and baseline visits as judged by the investigator
* Subjects with or without riluzole and/or edaravone. If using riluzole (any daily dose up to 100 mg), the dose must have been stable for at least 4 weeks before the screening visit and should not be changed during the study. If using edaravone, the treatment should have been started at least 4 weeks before the screening visit (at least one 28-day treatment cycle as indicated) and should not be changed during the study. If not on riluzole and/or edaravone, the respective treatments should not be started during the study

Exclusion Criteria:

* Subject in whom other causes of neuromuscular weakness have not been excluded
* Subject with a diagnosis of another neurodegenerative disease (e.g. Parkinson's or Alzheimer's disease)
* Assisted ventilation of any type within 3 months before the screening visit or at screening
* Any use of a diaphragm pacing system (DPS) within 3 months before the screening visit
* Any form of stem cell or gene therapy for the treatment of ALS
* Known hypersensitivity to levosimendan
* Administration of levosimendan within 3 months before the screening visit or previous participation in the present phase III study or earlier study with oral levosimendan in ALS patients (LEVALS)
* Any use of tirasemtiv or reldesemtiv within 1 month before the screening visit.
* Participation in a clinical trial with any experimental treatment within 30 days or within 5 half-lives of that treatment (whichever is longer) before the screening visit
* Any botulinum toxin use within 3 months before the screening visit
* Recorded diagnosis or evidence of major psychiatric diagnosis, significant cognitive impairment or clinically evident dementia that may interfere with the patient's ability to comply with study procedures
* Pulmonary illness (e.g. asthma or COPD) requiring regular treatment
* Haemodynamically significant uncorrected valve disease or hypertrophic cardiomyopathy or restrictive cardiomyopathy
* Any cardiovascular event (e.g. myocardial infarction, HF, arrhythmia or stroke) requiring hospitalisation within 3 months before the screening visit
* History of Torsades de Pointes (TdP) or diagnosed long QT-syndrome
* History of life-threatening ventricular arrhythmia, unless treated with reliable measures to prevent recurrence (e.g. with placement of implantable cardioverter defibrillator [ICD] or catheter ablation)
* History of second or third degree atrioventricular (AV) block or sinus node disease at screening, if not treated with pacemaker
* HR repeatedly > 100 bpm in the 12-lead ECG after a 5-minute rest at screening. If the HR is > 100 bpm in the first recording, then the second recording must be done after another 5 min rest to confirm HR > 100 bpm
* Systolic blood pressure (SBP) < 90 mmHg at screening
* Potassium < 3.7 mmol/l or > 5.5 mmol/l at screening
* Severe renal impairment (creatinine clearance < 30 ml/min at screening), creatinine > 170 μmol/l at screening or on dialysis
* Blood haemoglobin < 10 g/dl at screening or blood donation or loss of significant amount of blood within 60 days before the screening visit
* Clinically significant hepatic impairment at the discretion of the investigator
* Body mass index (BMI) ≤ 18.5kg/m2 (BMI = weight/height2)
* Women who are lactating or of reproductive age without a negative pregnancy test and without a commitment to using a highly effective method of contraception (e.g. oral hormonal contraceptives associated with inhibition of ovulation, intrauterine devices and long acting progestin agents), if sexually active during the study, and for 1 month after the last dose of the study treatment. Women who are postmenopausal (1 year since last menstrual cycle), surgically sterilised or who have undergone a hysterectomy are considered not to be reproductive and can be included
* Patient judged to be actively suicidal by the investigator during 3 months before the screening visit
* Patients with known history of human immunodeficiency virus (HIV) infection
* Any other clinically significant cardiovascular, gastrointestinal, hepatic, renal, neurological or psychiatric disorder or any other major concurrent illness that in the opinion of the investigator could interfere with the interpretation of the study results or constitute a health risk for the subject if he/she took part in the study

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 496 (Actual)
Dates: Start 2018-06-21 (Actual); Primary Completion 2020-07-23 (Actual); Study Completion 2020-07-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Merja Mäkitalo, CSD, Study Director — Orion Corporation, Orion Pharma
Locations (104):
- United States (48):
  - Phoenix Neurological Associates, Phoenix, Arizona
  - Neuromuscular Research Center and Neuromuscular Clinic of Arizona, Phoenix, Arizona
  - University of California San Diego, La Jolla, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - University of California Irvine, Orange, California
  - California Pacific Medical Center, San Francisco, California
  - Colorado Springs Neurological Associates, Colorado Springs, Colorado
  - Hospital for Special Care, New Britain, Connecticut
  - Georgetown University, Washington D.C., District of Columbia
  - The George Washington Medical Faculty Associates - Foggy Bottom North Pavilion, Washington D.C., District of Columbia
  - Providence Holy Cross Medical Center, Fort Lauderdale, Florida
  - University of Florida, Gainesville, Florida
  - University of Florida Health - Jacksonville, Jacksonville, Florida
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - University of South Florida, Tampa, Florida
  - Emory University School of Medicine, Atlanta, Georgia
  - Augusta University, Augusta, Georgia
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - University of Kentucky Chandler Medical Center, Lexington, Kentucky
  - Kentucky Neuroscience Research, Louisville, Kentucky
  - The Johns Hopkins Hospital, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - HealthPartners Specialty Center, Saint Paul, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Neurology Associates, Lincoln, Nebraska
  - Mount Sinai Beth Israel, New York, New York
  - Hospital for Special Surgery, New York, New York
  - Columbia Presbyterian Hospital, New York, New York
  - Neurosciences Institute - Neurology Charlotte, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - The Ohio State University, Columbus, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Providence Brain and Spine Institute, Portland, Oregon
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Temple University School of Medicine, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Texas Neurology, Dallas, Texas
  - Nerve and Muscle Center of Texas, Houston, Texas
  - University of Utah - Imaging & Neurosciences Center, Salt Lake City, Utah
  - University of Vermont Medical Center, Burlington, Vermont
  - Swedish Neuroscience Institute, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington
  - Froedtert Hospital, Milwaukee, Wisconsin
- Australia (5):
  - Brain and Mind Centre, Camperdown, New South Wales
  - Royal Brisbane and Women's Hospital, Brisbane, Queensland
  - Flinders Medical Centre, Bedford Park, South Australia
  - Calvary Health Care Bethlehem, Caulfield South, Victoria
  - Perron Institute for Neurological and Translational Science, Murdoch, Western Australia
- Austria (3):
  - Universität Innsbruck, Innsbruck, Tyrol
  - Salzkammergut-Klinikum Vöcklabruck, Vöcklabruck, Upper Austria
  - Medizinische Universität Wien, Vienna
- Belgium (3):
  - Universitaire Ziekenhuis Leuven, Leuven, Flemish Brabant
  - Centre Hospitalier Régional de la Citadelle, Liège, Liege
  - Algemeen Ziekenhuis St. Lucas Gent, Ghent, Oost-Vlaanderen
- Canada (9):
  - Alberta Health Services - Neuromuscular Clinic, Calgary, Alberta
  - University of Alberta, Edmonton, Alberta
  - Stan Cassidy Centre for Rehabilitation, Fredericton, New Brunswick
  - Moncton Hospital, Southeast Regional Health Authority, Moncton, New Brunswick
  - McMaster University Medical Centre, Hamilton, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Centre De Recherche Du Centre Hospitalier de l'Universite de Montreal - Hopital Notre-Dame, Montreal, Quebec
  - Montreal Neurological Institute and Hospital, Montreal, Quebec
  - Centre Hospitalier Affilie Universitaire de Quebec, Québec, Quebec
- Finland (3):
  - Neurologian Poliklinikka - Meilahden Tornisairaala 3, Helsinki
  - Etelä-Karjalan keskussairaala, Lappeenranta
  - Turku University Hospital, Turku
- France (4):
  - Centre Hospitalier Universitaire de Limoges, Limoges
  - Hôpital Gui de Chauliac, Montpellier
  - Hôpital Pasteur, Nice
  - Centre Hospitalier Régional et Universitaire de Tours Hôpital Bretonneau, Tours
- Germany (9):
  - Universitätsklinikum Ulm, Ulm, Baden-Wurttemberg
  - Deutsche Klinik für Diagnostik, Wiesbaden, Hesse
  - Medizinische Hochschule Hannover, Hanover, Lower Saxony
  - Universitätsmedizin Rostock, Rostock, Mecklenburg-western-pommerania
  - Alfried Krupp Krankenhaus Rüttenscheid, Essen, North Rhine-Westphalia
  - Universitätsklinikum Münster, Münster, North Rhine-Westphalia
  - Universitätsklinikum Carl Gustav Carus, Dresden, Saxony
  - Universitätsklinikum Jena, Jena, Thuringia
  - Charité Universitätsmedizin Berlin - Campus Virchow-Klinikum, Berlin
- Beaumont Hospital - Ireland, Dublin, Ireland
- Italy (6):
  - Azienda Ospedaliera Universitaria San Martino, Genova
  - Azienda Ospedaliera Universitaria-Maggiore della Carità di Novara, Novara
  - ICS Maugeri Spa SB, Pavia
  - Azienda Ospedaliero-Universitaria Pisana Ospedale Santa Chiara, Pisa
  - Policlinico Umberto I di Roma, Roma
  - Azienda Ospedaliera - Universitaria Città della Salute e della Scienza di Torino, Torino
- Netherlands (2):
  - Academisch Medisch Centrum, Amsterdam, North Holland
  - Universitair Medisch Centrum Utrecht - Rudolf Magnus Instituut voor Neurowetenschappen, Utrecht
- Spain (5):
  - Hospital de Basurto, Bilbao, Vizcaya
  - Hospital Universitari de Bellvitge, Barcelona
  - Hospital Universitario Reina Sofia, Córdoba
  - Hospital San Rafael - Madrid, Madrid
  - Hospital Universitario y Politécnico de La Fe, Valencia
- Sweden (3):
  - Norrlands Universitetssjukhus, Umeå, Västerbotten County
  - Centralsjukhuset Karlstad, Karlstad
  - Karolinska Universitetssjukhuset, Stockholm
- United Kingdom (3):
  - Barts Health NHS Trust, London, England
  - King's College Hospital NHS Foundation Trust, London, England
  - The Walton Centre NHS Foundation Trust, Liverpool

REFERENCES:
- [Derived] Cudkowicz M, Genge A, Maragakis N, Petri S, van den Berg L, Aho VV, Sarapohja T, Kuoppamaki M, Garratt C, Al-Chalabi A; REFALS investigators. Safety and efficacy of oral levosimendan in people with amyotrophic lateral sclerosis (the REFALS study): a randomised, double-blind, placebo-controlled phase 3 trial. Lancet Neurol. 2021 Oct;20(10):821-831. doi: 10.1016/S1474-4422(21)00242-8. PMID 34536404

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with amyotrophic lateral sclerosis (ALS) were recruited.
Pre-assignment Details: Male or female subjects with a diagnosis of probable or definite ALS according to El Escorial revised criteria, disease duration from symptom onset of 12-48 months, written or verbal IC obtained. Able to swallow study treatment capsules. Sitting SVC between 60-90% of the predicted value at screening visit. Stable riluzole and/or edaravone allowed.
Period: Overall Study
Arm/Group | Levosimendan | Placebo for Levosimendan
Started | 329 | 167
Completed | 217 | 112
Not Completed | 112 | 55
Not completed — Protocol Violation | 1 | 0
Not completed — Death | 9 | 8
Not completed — Consent withdrawn by subject | 6 | 1
Not completed — Lost to Follow-up | 5 | 3
Not completed — Adverse Event | 26 | 9
Not completed — Disease progression | 33 | 17
Not completed — Other | 11 | 5
Not completed — Personal reason | 21 | 12

BASELINE CHARACTERISTICS:
Population: Intention-to-treat (ITT) dataset, including all randomised subjects, was used for the primary evaluation. Sensitivity analyses using full analysis set (FAS) and two per-protocol (PP) datasets (up to 12 weeks and up to 48 weeks) were performed. FAS included all treated subjects with at least one post baseline SVC measurement. PP dataset included all randomised subjects except subjects with relevant major protocol deviations.
Groups:
- Total: Total of all reporting groups
Arm/Group | Levosimendan | Placebo for Levosimendan | Total
Number analyzed (Participants) | 329 | 167 | 496
Age, Continuous [Mean (Standard Deviation); unit: years] | 59 (11.2) | 59.7 (10.8) | 59.3 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 122 | 67 | 189
  Male | 207 | 100 | 307
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 9 | 1 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 3 | 8
  White | 305 | 157 | 462
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 9 | 6 | 15
Region of Enrollment [Number; unit: participants]
  United States | 105 | 45 | 150
  United Kingdom | 8 | 1 | 9
  Spain | 44 | 15 | 59
  Canada | 25 | 22 | 47
  Austria | 6 | 1 | 7
  Netherlands | 8 | 8 | 16
  Sweden | 19 | 7 | 26
  Belgium | 12 | 10 | 22
  Ireland | 3 | 2 | 5
  Finland | 10 | 3 | 13
  Italy | 18 | 16 | 34
  Australia | 14 | 6 | 20
  France | 3 | 5 | 8
  Germany | 54 | 26 | 80

OUTCOME MEASURES:

1. Primary Outcome: Supine Slow Vital Capacity (SVC)
Description: Change from baseline to 12 weeks, expressed as % of predicted normal.
Time Frame: The change from baseline at 12 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage
Arm/Group | Levosimendan | Placebo for Levosimendan
Number analyzed (Participants) | 329 | 167
percentage | -6.731 [-8.290 to -5.171] | -6.988 [-9.052 to -4.925]
Statistical Analysis 1: Comparison: Levosimendan vs Placebo for Levosimendan; Test type: Superiority; p = 0.8253, ANCOVA; Mean Difference (Final Values) = 0.258, 95% CI 2-sided [-2.032 to 2.547]

2. Secondary Outcome: Combined Assessment of Function and Survival Through 48 Weeks
Description: Scale: The ALS Functional Rating Scale - Revised. This scale includes 12 items. Each item was scored from 0 to 4. Total score is the sum of the scores of all 12 items. Each subject is ranked according to time-to-death (earlier deaths ranked lower than later deaths). Subjects who survive are ranked more favorably than subjects who died. Among the survivors, subjects are ranked according to change in ALSFRS-R (greater worsening of ALSFRS-R is ranked lower than after deaths). Subjects who survive are ranked more favorably than subjects who died. Among the survivors, subjects are ranked according to change in ALSFRS-R (greater worsening of ALSFRS-R is ranked lower than less worsening or an improvement in ALSFRS-R). The ranked scores range from 001 to 496 (the number of participants assessed for the Outcome Measure) with larger rank score numbers associated with a better outcome.
Time Frame: Mean rank at 48 weeks
Measure: Least Squares Mean (Standard Error); unit: Scores on a rank scale
Arm/Group | Levosimendan | Placebo for Levosimendan
Number analyzed (Participants) | 329 | 167
Scores on a rank scale | 239.85 (10.98) | 229.16 (13.31)
Statistical Analysis 1: Comparison: Levosimendan vs Placebo for Levosimendan; Test type: Superiority; p = 0.4277, ANCOVA; Mean Difference (Final Values) = 10.69, 95% CI 2-sided [-15.74 to 37.12]

3. Secondary Outcome: Time to Respiratory Event Through 48 Weeks
Description: ALSFRS-R scale contains 3 items that relate to respiratory function: severity of dyspnoea, occurrence of orthopnoea (shortness of breath when lying flat) and the use of mechanical ventilation for respiratory insufficiency. A reduction in any one of these items was considered a respiratory event. Not all patients receive ventilatory support, despite respiratory insufficiency: meeting "protocolised" criteria for NIV relates to patients without NIV whose slow vital capacity declined to a level that would ordinarily trigger such treatment.
Time Frame: Time to event through 48 weeks
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Levosimendan | Placebo for Levosimendan
Number analyzed (Participants) | 329 | 167
Days | 90 [82 to 144] | 126 [82 to 169]
Statistical Analysis 1: Comparison: Levosimendan vs Placebo for Levosimendan; Test type: Superiority; p = 0.6733, Regression, Cox; Hazard Ratio (HR) = 1.051, 95% CI 2-sided [0.833 to 1.327]

4. Secondary Outcome: Change From the Baseline in Clinical Global Impression CGI at 48 Weeks
Description: Visual Analogue Scale 0-100 millimeters, rated by study subjects. Score 0 indicates that the subject is completely well without any disability and score 100 indicates the worst possible severity of the condition.
Time Frame: The change from baseline at 48 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Levosimendan | Placebo for Levosimendan
Number analyzed (Participants) | 329 | 167
units on a scale | 17.048 [14.111 to 19.984] | 13.285 [9.252 to 17.318]
Statistical Analysis 1: Comparison: Levosimendan vs Placebo for Levosimendan; Test type: Superiority; p = 0.1295, ANCOVA; Mean Difference (Final Values) = 3.762, 95% CI 2-sided [-1.129 to 8.654]

5. Secondary Outcome: Change From Baseline in Respiratory Function of ALSFRS-R at 48 Weeks
Description: ALSFRS-R scale contains 3 items that relate to respiratory function: severity of dyspnoea, occurrence of orthopnoea (shortness of breath when lying flat) and the use of mechanical ventilation for respiratory insufficiency. These are added together to created the respiratory domain with a score range 0-12 (where 12 represents normal function). Although individual items and patients vary, ALSFRS-R typically declines at a relatively constant rate over time. Plotted over time the slope of the line obtained indicates the speed of progression and thus an effective treatment might be expected to reduce the slope of decline.
Time Frame: Slope of decline at 48 weeks
Measure: Least Squares Mean (Standard Error); unit: Score on a scale/month
Arm/Group | Levosimendan | Placebo for Levosimendan
Number analyzed (Participants) | 329 | 167
Score on a scale/month | -0.191 (0.015) | -0.205 (0.022)
Statistical Analysis 1: Comparison: Levosimendan vs Placebo for Levosimendan; Test type: Superiority; p = 0.6230, Mixed Models Analysis; Mean Difference (Final Values) = 0.013, 95% CI 2-sided [-0.040 to 0.066]

6. Secondary Outcome: Supine Borg Category Ratio 10 Scale at 12 Weeks
Description: Patients rated their perception of the severity of their dysnoea using the Borg scale. The scale ranges from 0 (no dyspnoea) to 10 (maximal). Each category is numbered and most (not all) have verbal cues. At each assessment the patient scored the category they felt best described their symptoms. The analysis measured change from baseline at 12 weeks, where a negative score indicates improvement and a positive score reflects worsening.
Time Frame: Change from baseline at 12 weeks
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Levosimendan | Placebo for Levosimendan
Number analyzed (Participants) | 329 | 167
score on a scale | -0.152 (0.138) | 0.120 (0.186)
Statistical Analysis 1: Comparison: Levosimendan vs Placebo for Levosimendan; Test type: Superiority; p = 0.1752, ANCOVA; Mean Difference (Final Values) = -0.272, 95% CI 2-sided [-0.666 to 0.122]

ADVERSE EVENTS:
Time Frame: From signing an informed consent until 25 days from stopping the treatment, up to 51 weeks.
Description: Four randomised patients - three in the levosimendan group and one in the placebo group - did not start study treatment and so are not included in the safety population.
Arm/Group | Levosimendan | Placebo for Levosimendan
All-Cause Mortality (participants affected / at risk) | 27/326 | 17/166
Serious Adverse Events (participants affected / at risk) | 89/326 | 45/166
Other Adverse Events (participants affected / at risk) | 312/326 | 157/166
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Levosimendan (N=326) | Placebo for Levosimendan (N=166)
Breast cancer (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Hypopharyngeal cancer (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Invasive ductal breast carcinoma (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Metastases to liver (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac arrest (Cardiac disorders) | 2 (2) | 1 (1)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 2 (2) | 0 (0)
Coronary artery dissection (Cardiac disorders) | 0 (0) | 1 (1)
Diastolic dysfunction (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 3 (3) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Stress cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 2 (2) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Hypertrophic cardiomyopathy (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Vertigo positional (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric ulcer hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 2 (2) | 0 (0)
Ileus paralytic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Peptic ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0)
Cardiac death (General disorders) | 0 (0) | 1 (1)
Catheter site inflammation (General disorders) | 1 (2) | 0 (0)
Chest pain (General disorders) | 4 (4) | 1 (1)
Death (General disorders) | 0 (0) | 1 (1)
Euthanasia (General disorders) | 1 (1) | 0 (0)
Sudden death (General disorders) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Catheter site cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Catheter site infection (Infections and infestations) | 1 (1) | 1 (1)
Enterobacter bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 12 (12) | 7 (10)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 0 (0)
Pulmonary sepsis (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 1 (1)
Septic shock (Infections and infestations) | 1 (1) | 0 (0)
Serratia bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Stoma site infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 5 (5)
Urinary tract infection bacterial (Infections and infestations) | 1 (1) | 0 (0)
Vascular device infection (Infections and infestations) | 1 (1) | 0 (0)
Brain contusion (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Facial bones fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 13 (13) | 6 (7)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lip injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural hemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Skull fractured base (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Ulna fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Amyotrophic lateral sclerosis (Nervous system disorders) | 4 (4) | 3 (3)
Brain injury (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 3 (3) | 0 (0)
Hypercapnic coma (Nervous system disorders) | 1 (1) | 0 (0)
Intraventricular haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Lacunar stroke (Nervous system disorders) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 1 (1) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 2 (2) | 0 (0)
Unresponsive to stimuli (Nervous system disorders) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (1) | 2 (2)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Restlessness (Psychiatric disorders) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Neurogenic bladder (Renal and urinary disorders) | 1 (1) | 0 (0)
Urethral obstruction (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 2 (2) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 3 (4)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Hypoventilation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 8 (9) | 2 (2)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 4 (4)
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory depression (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 13 (13) | 5 (5)
Respiratory muscle weakness (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Aortic stenosis (Vascular disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 2 (2) | 1 (1)
Hypertensive crisis (Vascular disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 2 (2) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Levosimendan (N=326) | Placebo for Levosimendan (N=166)
Palpitations (Cardiac disorders) | 17 (23) | 4 (4)
Sinus tachycardia (Cardiac disorders) | 13 (14) | 0 (0)
Tachycardia (Cardiac disorders) | 32 (41) | 8 (11)
Abdominal pain (Gastrointestinal disorders) | 12 (13) | 2 (2)
Constipation (Gastrointestinal disorders) | 38 (41) | 21 (22)
Diarrhoea (Gastrointestinal disorders) | 26 (31) | 14 (18)
Dysphagia (Gastrointestinal disorders) | 47 (55) | 27 (31)
Nausea (Gastrointestinal disorders) | 29 (35) | 15 (17)
Salivary hypersecretion (Gastrointestinal disorders) | 22 (23) | 9 (10)
Asthenia (General disorders) | 16 (19) | 1 (1)
Fatigue (General disorders) | 30 (33) | 10 (11)
Oedema peripheral (General disorders) | 26 (28) | 12 (14)
Nasopharyngitis (Infections and infestations) | 52 (62) | 26 (31)
Upper respiratory tract infection (Infections and infestations) | 13 (16) | 5 (5)
Urinary tract infection (Infections and infestations) | 25 (31) | 17 (22)
Heart rate increased (Investigations) | 64 (68) | 5 (5)
Weight decreased (Investigations) | 26 (27) | 15 (15)
Contusion (Injury, poisoning and procedural complications) | 21 (23) | 8 (9)
Fall (Injury, poisoning and procedural complications) | 86 (150) | 45 (100)
Skin laceration (Injury, poisoning and procedural complications) | 17 (20) | 12 (15)
Arthralgia (Musculoskeletal and connective tissue disorders) | 13 (15) | 9 (9)
Back pain (Musculoskeletal and connective tissue disorders) | 14 (16) | 7 (11)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 17 (21) | 7 (8)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 31 (39) | 18 (18)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 14 (17) | 8 (8)
Neck pain (Musculoskeletal and connective tissue disorders) | 10 (11) | 6 (6)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 24 (28) | 6 (6)
Dizziness (Nervous system disorders) | 21 (35) | 13 (14)
Headache (Nervous system disorders) | 101 (142) | 36 (49)
Anxiety (Psychiatric disorders) | 18 (18) | 6 (6)
Depression (Psychiatric disorders) | 13 (13) | 4 (4)
Insomnia (Psychiatric disorders) | 22 (22) | 10 (10)
Cough (Respiratory, thoracic and mediastinal disorders) | 16 (19) | 13 (15)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 54 (61) | 30 (35)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 17 (17) | 12 (12)
Hypertension (Vascular disorders) | 8 (8) | 9 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-03-26): https://cdn.clinicaltrials.gov/large-docs/21/NCT03505021/Prot_000.pdf
  • Statistical Analysis Plan (2020-06-18): https://cdn.clinicaltrials.gov/large-docs/21/NCT03505021/SAP_001.pdf